CLINICAL TRIAL: NCT05099887
Title: Use of Procenta® Conformable Barrier in Recovery of Non-Healing Foot & Ankle Ulcers in Patients With Diabetes Mellitus Types I and II
Brief Title: Use of Procenta® Conformable Barrier for Non-Healing Foot & Ankle Ulcers in Patients With Diabetes Mellitus Types I and II
Acronym: Procenta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The VA Western New York Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1591772
Record Dates: First submitted 2021-05-17; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- wound application (Other): Application of Procenta as wound cover
  Interventions: Biological: Procenta conformable barrier

INTERVENTIONS:
Biological: Procenta conformable barrier — Wound care dressing biologic allograft

SUMMARY:
Procenta® has been successful in facilitating closure of non-healing diabetic ulcers in patients where proper wound care management/practice has failed along with other allo- and xenografts. In each individual case study where diabetes mellitus was pathological, unique wound morphologies with high variability in all three dimensions showed significant progress or were fully closed after at least one application of Procenta®. In the present study, the investigators seek to investigate the efficacy of the product over a 90-day treatment time-course with a larger sample size of patients suffering from non-healing wounds due to diabetes mellitus types I or II (diabetes mellitus). As a result, the investigators hope to better understand the potential and limitations of the product under these conditions with the anticipation that a significant number of patients will recover, avoid amputation, and return to a normal daily life.

DETAILED DESCRIPTION:
Study Design Overview:

Potential candidates are diabetes mellitus type I or II patients with ulcers on the foot and ankle with no-to-minimal associated co-morbidities, regardless of age. The investigators anticipate the patient pool is likely to be in the range of 60-95 years of age. For this study, patients must have failed previous treatments which are in accordance with proper wound management practices and are considered to be typical applications/regiments. Patient's eligible for the current study should be candidates for amputation and failed traditional wound care practices and treatment alternatives. Diabetic ulcers of the foot and ankle should have a minimum surface area of 0.5cm2 and a maximum of 10.0 cm2.

Patients meeting selection criteria should be consulted regarding the application of Procenta® as an alternative to other treatments and/to surgeries. Once properly advised, the patient enrollment will begin with the execution of the Research Informed Consent Document from the Department of Veterans Affairs and the document, Informed Consent for Use of Procenta® for VAWNY072020PRODFU (IRB693) for the study. When scheduled for Procenta® application, the physician will complete form, Initial Application Form for VAWNY072020PRODFU (IRB692.F02), where the condition of the ulcer and procedure data will be recorded.

Application of one unit of the tissue allograft Procenta® (Catalog # 001050, 200mg) per ≤2.5cm2 ulcer surface area will be the protocol standard. Up to 4 units may be applied to a wound within the range described at each office visit and should fill ≥70% of the wound volume. The study will enroll 10 patients, where Procenta® is applied up to once every 7 days over a 12-week time-course. Data will be collected in the form of physician reporting during the initial application and at each follow-up visit on forms, Initial Application Form for VAWNY072020PRODFU (IRB692.F02) and Week (1-12) Follow-Up Form for VAWNY072020PRODFU (IRB692.F03). The patient will also be required to report on their quality of life at each follow-up on the Quality of Life Questionnaire for VAWNY072020PRODFU (IRB692.F04) and Foot and Ankle Ability Measure (FAAM) at the time of enrollment and at the end of the study period. Patients must agree to a 90-day treatment period, as well as a standard 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Patient must have a non-healing ulcer associated with diabetes mellitus
  * Ulcer must have a minimum surface area of 0.5cm2 and a maximum surface area of 10.0cm2 i. Wound depth is not a criterion, though it will be documented throughout the study
  * Failed conventional wound care treatments
  * Amputation candidate

Exclusion Criteria:

* Exclusion Criteria:

  * Co-morbidities which do not allow the ulcer to be linked to diabetic pathology will be excluded from the study

    o This is intended to limit the number of probable causes/contributing factors related to the ulcer. Commonly associated conditions, such as peripheral vascular disease is not an exclusion criterion, though it is documented in form, Enrollment Application Form for VAWNY072020PRODFU (IRB692.F01)
  * Wounds with active infections or gangrene
  * Active carcinoma(s)
  * Wounds where bone is necrosing, avascular necrosis
  * Multiple ulcers on the same foot/ankle

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent of Wound closure | through study completion, approximately 6 months
  Primary end points are percent of wound closure

IPD SHARING:
Plan to Share IPD: No